CLINICAL TRIAL: NCT01382992
Title: A Retrospective EGFR Mutation Status Study in Chinese NSCLC Patients Using Paired Plasma and Tissue Samples
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Mengzhao Wang, Peking Union Medical College Hospital
Other Study IDs: LCC001
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; erbB-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin-fixed, paraffin-embedded tissue slices and plasma samples are to be retained.

GROUPS / COHORTS (2):
- Early Stage
- Late Stage

SUMMARY:
EGFR mutations plays an essential role in EGFR-TKIs treatment. However, for some patients, tissue samples are not available. The purpose of this study is to determine whether blood sample is feasible for EGFR mutation detection.For late stage NSCLC, we hypothesis plasma sample is an alternative for detecting EGFR mutations.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer
* Available plasma and pathologically confirmed tissue slices(pre-chemo and pre-radio therapy)
* Informed Consent

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients who were diagnosed or treated in Peking Union Medical College Hospital or Peking University People's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-06

PRIMARY OUTCOMES:
To determine the consistence of EGFR mutation status in paired tissue and plasma samples | 3 months

SECONDARY OUTCOMES:
To determine the EGFR mutation status in Chinese NSCLC | 3month

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China